CLINICAL TRIAL: NCT07061691
Title: WIM Exosuit Wearable Soft Robot for Enhancing Walking Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator:Arun Jayaraman, PT, PhD,Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00221889
Record Dates: First submitted 2025-06-27; First posted 2025-07-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Healthy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Population (Experimental)
  Interventions: Device: WIM Robotic Exoskeleton

INTERVENTIONS:
Device: WIM Robotic Exoskeleton — Wearable hip-powered exoskeleton

SUMMARY:
This study is to develop, test, and optimize a soft hip wearable robot for individuals who have experience a stroke.

ELIGIBILITY:
Inclusion Criteria:

* - Be at least 6 months post-stroke, have a diagnosis of Parkinson's, have a diagnosis of multiple sclerosis, or an adult older than 65 with no known neurological diagnoses.

For the Optimization Aim of the study, Participants may also be healthy individuals with no known impairments.

* Age: 18-89 years of age
* For stroke, Parkinson's, multiple sclerosis, or older adult participants, must have adequate cognitive function (MMSE score >17)
* Ability to walk at least 10 meters with maximum of 1 person assist
* Able to safely fit into the WIM exosuit, which is confirmed via an in-person fitting..

Exclusion Criteria:

* - <90 days post major orthopedic surgery (i.e. hip, knee, and/or ankle joint replacement.)
* < 6 months post CABG or cardiac valve procedure
* Any skin irritations / conditions that may preclude a participant from tolerating the use of the exosuit.
* Severe osteoporosis, defined as osteoporosis that has been diagnosed and a participant's doctor has recommended pharmacologic treatment, or there is both a history of osteoporosis and a history of fractures.
* Serious cardiac conditions, such as hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living.
* Pregnancy
* Uncontrolled hypertension (resting systolic blood pressure greater than or equal to 150, or resting diastolic pressure greater than or equal to 90.) If a participant demonstrates a BP greater than these values, then the participant will sit quietly for 5 mins, and then be re-checked. If the BP values remain over those thresholds, then the participant will be excluded. Individuals in such situations may return to be re-screened for participation after they follow up with their physician and the hypertension is better controlled.
* Lower extremity fracture, either currently or within the past 6 months.
* Modified Ashworth Spasticity (MAS) scores of ≥ 3 in hip flexors or extensors, if the participant is post-stroke or multiple sclerosis.
* Pre-existing neurological disorders such as amyotrophic lateral sclerosis (ALS), dementia
* History of major head trauma, lower extremity amputation, non-healing ulcers of a lower extremity, ongoing active infections, legal blindness, or a history of significant psychiatric illness.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | Baseline (Single-session)
  Primary outcome for Optimization aim of study.
Metabolic Cost | Baseline (single session)
  Primary outcome for Optimization aim of study. Data collected using Cosmed K5 Metabolic Unit

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No